CLINICAL TRIAL: NCT03168321
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2 Arm, Parallel Group Study Comparing the Safety and Efficacy of IDP-123 Lotion and IDP-123 Vehicle Lotion in the Treatment of Acne Vulgaris
Brief Title: A Phase 3, Vehicle-controlled Efficacy and Safety Study of IDP-123 Lotion in the Treatment of Acne Vulgaris (301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V01-123A-301
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-123 Lotion (Experimental): Tazarotene 0.045% Lotion
  Interventions: Drug: IDP-123 Lotion
- IDP-123 Vehicle Lotion (Placebo Comparator): Vehicle Lotion
  Interventions: Drug: IDP-123 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-123 Lotion — Tazarotene 0.045% Lotion
  Other Names: IDP-123
  Arms: IDP-123 Lotion
Drug: IDP-123 Vehicle Lotion — Vehicle Lotion
  Other Names: Vehicle
  Arms: IDP-123 Vehicle Lotion

SUMMARY:
This is a multicenter, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, efficacy, and tolerability of IDP-123 Lotion in comparison with IDP-123 Vehicle Lotion.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, efficacy, and tolerability of IDP-123 Lotion and IDP-123 Vehicle Lotion. To be eligible for the study subjects must be at least 9 years of age and have a clinical diagnosis of moderate to severe acne.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 9 years of age and older;
2. Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit);
3. Subject must have a score of 3 (moderate) or 4 (severe) on the Evaluator's Global Severity assessment at the baseline visit;
4. Subjects with facial acne inflammatory lesion (papules, pustules, and nodules) count no less than 20 but no more than 50;
5. Subjects with facial acne non-inflammatory lesion (open and closed comedones) count no less than 25 but no more than 100;
6. Subjects with two or fewer nodules

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study;
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram-negative folliculitis, dermatitis, eczema;
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive;
4. Subjects with a facial beard or mustache that could interfere with the study assessments;
5. Subjects with more than two (2) facial nodules;
6. Evidence or history of cosmetic-related acne

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (45):
- United States (42):
  - Valeant Site 19, Phoenix, Arizona
  - Valeant Site 21, Phoenix, Arizona
  - Valeant Site 24, Hot Springs, Arkansas
  - Valeant Site 04, La Mesa, California
  - Valeant Site 02, Manhattan Beach, California
  - Valeant Site 42, Murrieta, California
  - Valeant Site 39, Sacramento, California
  - Valeant Site 01, San Diego, California
  - Valeant Site 37, Wheat Ridge, Colorado
  - Valeant Site 35, Boca Raton, Florida
  - Valeant Site 40, North Miami Beach, Florida
  - Valeant Site 33, Ormond Beach, Florida
  - Valeant Site 27, Pembroke Pines, Florida
  - Valeant Site 13, Sanford, Florida
  - Valeant Site 03, West Palm Beach, Florida
  - Valeant Site 26, Newnan, Georgia
  - Valeant Site 30, Boise, Idaho
  - Valeant Site 06, Arlington Heights, Illinois
  - Valeant Site 23, New Albany, Indiana
  - Valeant Site 17, South Bend, Indiana
  - Valeant Site 31, Overland Park, Kansas
  - Valeant Site 22, Louisville, Kentucky
  - Valeant Site 08, Metairie, Louisiana
  - Valeant Site 38, Detroit, Michigan
  - Valeant Site 16, Warren, Michigan
  - Valeant site 20, New York, New York
  - Valeant Site 36, New York, New York
  - Valeant Site 09, High Point, North Carolina
  - Valeant Site 32, Cincinnati, Ohio
  - Valeant Site 11, Dublin, Ohio
  - valeant Site 07, Gresham, Oregon
  - Valeant Site 15, Johnston, Rhode Island
  - Valeant Site 34, Knoxville, Tennessee
  - valeant Site 14, Nashville, Tennessee
  - Valeant Site 12, Austin, Texas
  - Valeant Site 05, Katy, Texas
  - Valeant Site 18, Plano, Texas
  - Valeant Site 25, San Antonio, Texas
  - Valeant Site 43, Webster, Texas
  - Valeant Site 41, Salt Lake City, Utah
  - Valeant Site 45, Norfolk, Virginia
  - Valeant Site 44, Spokane, Washington
- Canada (3):
  - Valeant Site 29, Peterborough, Ontario
  - Valeant Site 28, Waterloo, Ontario
  - Valeant Site 10, Laval, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- IDP-123 Lotion: IDP-123 (Tazarotene 0.045%) Lotion
- Vehicle Lotion: IDP-123 Vehicle Lotion
Period: Overall Study
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Started | 402 | 411
Completed | 347 | 356
Not Completed | 55 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-123 Lotion | Vehicle Lotion | Total
Number analyzed (Participants) | 402 | 411 | 813
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (7.29) | 20.4 (6.94) | 20.6 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 271 | 551
  Male | 122 | 140 | 262
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 15 | 13 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 76 | 83 | 159
  White | 293 | 297 | 590
  More than one race | 11 | 10 | 21
  Unknown or Not Reported | 4 | 3 | 7
Lesion counts [Mean (Standard Deviation); unit: lesions] — For noninflammatory facial lesions, open comedones (blackheads) and closed comedones (whiteheads) were recorded as a single count. For inflammatory facial lesions, papules (solid, elevated lesion less than 5 mm) and pustules (elevated lesion containing pus less than 5 mm) were recorded as a single count, while nodular lesions (palpable subcutaneous lesion greater than 5 mm) were counted and recorded separately.
  lesions
    Non-inflammatory lesions | 41.1 (15.67) | 40.7 (16.29) | 40.9 (15.98)
    Inflammatory lesions | 28.5 (7.04) | 28.1 (7.04) | 28.3 (7.04)
Evaluator's Global Severity Score [Count of Participants; unit: Participants] — Evaluator's Global Severity Score (EGSS) was determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations were scored on a scale of 0-4, with 0 being clear and 4 being severe.
  Participants
    Moderate | 368 | 384 | 752
    Severe | 34 | 27 | 61

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Lesion Counts at Week 12
Description: For noninflammatory facial lesions, open comedones (blackheads) and closed comedones (whiteheads) were recorded as a single count. For inflammatory facial lesions, papules (solid, elevated lesion less than 5 mm) and pustules (elevated lesion containing pus less than 5 mm) were recorded as a single count, while nodular lesions (palpable subcutaneous lesion greater than 5 mm) were counted and recorded separately.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: lesion counts
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 402 | 411
lesion counts
  Non-inflammatory lesions | -21.0 (14.72) | -16.4 (14.52)
  Inflammatory lesions | -15.6 (10.41) | -12.4 (10.43)

2. Primary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS) and Had an EGSS at Week 12 That Equated to "Clear" or "Almost Clear"
Description: Evaluator's Global Severity Score (EGSS) was determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations were scored on a scale of 0-4, with 0 being clear and 4 being severe.
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 402 | 411
percentage of participants | 25.5 | 13.0

3. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 12
Description: as for outcome 1
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 402 | 411
percentage change
  Non-inflammatory lesions | -51.36 (36.397) | 41.47 (35.223)
  Inflammatory lesions | -55.52 (36.531) | -45.70 (36.984)

4. Secondary Outcome: Percentage of Subjects Who Had at Least a 2-grade Reduction From Baseline at Week 12 in the Evaluator's Global Severity Score (EGSS)
Description: as for outcome 2
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 402 | 411
percentage of participants | 28.3 | 15.2

5. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 8
Description: as for outcome 1
Time Frame: Baseline to Week 8
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 402 | 411
percentage change
  Non-inflammatory lesions | -43.08 (32.430) | -34.34 (31.684)
  Inflammatory lesions | -45.30 (34.351) | -38.96 (34.548)

6. Secondary Outcome: Percentage Change in Mean Lesion Counts at Week 4
Description: as for outcome 1
Time Frame: Baseline to Week 4
Measure: Least Squares Mean (Standard Deviation); unit: percentage change
Arm/Group | IDP-123 Lotion | Vehicle Lotion
Number analyzed (Participants) | 402 | 411
percentage change
  Non-inflammatory lesions | -29.43 (32.441) | -23.25 (31.817)
  Inflammatory lesions | -27.27 (34.980) | -29.70 (34.368)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety population included all participants who received at least one confirmed dose of study drug and had at least one post-baseline safety assessment. There were 10 participants in the IDP-123 Lotion and 12 participants in the IDP-123 Vehicle Lotion group who did not have any post-baseline safety assessment.
Arm/Group | IDP-123 Lotion | Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/392 | 0/399
Serious Adverse Events (participants affected / at risk) | 3/392 | 3/399
Other Adverse Events (participants affected / at risk) | 0/392 | 0/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-123 Lotion (N=392) | Vehicle Lotion (N=399)
Abortion induced (Surgical and medical procedures) | 1 | 1
Abortion spontaneous (Surgical and medical procedures) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT03168321/Prot_SAP_000.pdf